CLINICAL TRIAL: NCT03364712
Title: Measurement of B Lymphocyte Stimulator (BLyS) in Peripheral Blood From Pregnant and Nonpregnant Women
Brief Title: Maternal Serum BLyS Levels Throughout Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, William Stohl, Professor of Medicine, University of Southern California
Other Study IDs: #HS-11-00449
Record Dates: First submitted 2017-10-16; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Pregnancy
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Banked sera.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant: Pregnant women receiving routine medical care, including venipuncture.
  Interventions: Other: routine medical care, venipuncture
- non-pregnant: Women not pregnant receiving routine medical care, including venipuncture.
  Interventions: Other: routine medical care, venipuncture

INTERVENTIONS:
Other: routine medical care, venipuncture

SUMMARY:
Background and rationale: B lymphocyte stimulator (BLyS) is a potent B cell survival factor that has been found to be elevated in patients with inflammatory conditions, such as systemic lupus and rheumatoid arthritis. Because of the immunologic changes associated with pregnancy, including changes in levels of T and B lymphocytes, it is postulated that BLyS levels would be altered in pregnancy compared to the non-pregnant state.

Objectives: The primary objective of this study is to assess the levels of BLyS in each trimester of pregnancy. Secondary objectives include evaluation of an association between BLyS levels and adverse pregnancy events; comparison of BLyS levels between healthy pregnant women and pregnant women with a medical or obstetric conditions; and, assessment of APRIL levels and comparison between APRIL levels and BLyS levels in study subjects.

Study population: Pregnant and non-pregnant women receiving care in the outpatient Obstetrics and Gynecology clinics at LAC+USC Medical Center.

Study methodology: Peripheral blood samples will be drawn from pregnant women and non-pregnant controls. Pregnant women will have blood drawn each trimester, at delivery, and postpartum, and control subjects will have blood drawn once, upon enrollment in the study.

Study outcomes: BLyS and APRIL levels during each trimester, postpartum and in cord blood will be compared between healthy pregnant women, pregnant women with a medical condition, and healthy non-pregnant controls. Additionally, pregnancy outcomes will be recorded to determine whether BLyS or APRIL levels correlate with adverse events.

Statistics: Continuous data will be analyzed by Student t-test or logistic regression, where appropriate. Categorical data will be analyzed using Chi square.

DETAILED DESCRIPTION:
The investigators performed a prospective observational study of pregnant women presenting for prenatal care at Los Angeles County+University of Southern California Obstetrics clinics. Subjects were recruited from October 2011 through June 2013. Pregnant women were recruited at the time of their first prenatal visit. Women under the age of 18 and women carrying a fetus with a known major congenital anomaly were excluded. A control group of premenopausal nonpregnant (NP) women without known medical or rheumatic illnesses was recruited from the Los Angeles County+University of Southern California Gynecology outpatient clinics. Informed consent was obtained from each study participant before enrollment. Approval for this study was obtained from the Los Angeles County+University of Southern California Institutional Review Board.

A participant was classified as having gestational hypertension if the participant had ≥2 episodes of new-onset HTN (systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg) after 20 weeks of pregnancy. PE was defined as gestational hypertension that was accompanied by proteinuria of at least 300 mg in a 24-hour urine collection or a protein/creatinine ratio ≥0.3. HELLP syndrome was diagnosed when a woman had laboratory evidence of hemolysis, a platelet count <100,000/μL, and serum levels of aspartate aminotransferase and alanine aminotransferase that were greater than or equal to twice normal values. Superimposed preeclampsia was diagnosed in a participant with CHTN when the participant experienced an acute exacerbation of hypertension after 20 weeks of gestation. In a participant without preexisting proteinuria, new-onset proteinuria was also required for the diagnosis.

Patient characteristics were obtained through patient interviews and medical chart review. Maternal venous blood was collected by venipuncture at least once per trimester, on admission for delivery, and postpartum. The first trimester was defined as <14 gestational weeks, the second trimester as 14 0/7 to 27 6/7 gestational weeks, and the third trimester as 28 0/7 gestational weeks to delivery. Postpartum samples were collected before hospital discharge after delivery.

Blood samples were collected in sterile tubes without additives and refrigerated until processing. Sera were routinely isolated from the clotted blood samples within 12 to 24 hours and were aliquotted and stored at -80°C. Serum BAFF levels were measured in a blinded fashion using a sandwich ELISA.

Chi-squared or Fisher exact testing was used for categorical variables, and Kruskal-Wallis or signed-ranks testing was used for all continuous variables. All tests were 2-sided, with a P value <0.05 considered statistically significant. Means are expressed as ± the SD. Medians are presented for data not normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman

Exclusion Criteria:

* Unable to give informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women seen at a single medical center
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
first-trimester serum blys level | up to 13 weeks of pregnancy (first trimester)
  maternal serum blys level during the first trimester of pregnancy
second-trimester serum blys level | from 14 through 26 weeks of pregnancy (second trimester)
  maternal serum blys level during the second trimester of pregnancy
third-trimester serum blys level | from 27 weeks of pregnancy through delivery of baby (third trimester of pregnancy)
  maternal serum blys level during the third trimester of pregnancy
cord blood serum blys level | delivery of baby
  serum blys level in cord blood obtained at delivery
post-partum serum blys level | 1-2 days post-partum
  maternal serum blys level post-partum